CLINICAL TRIAL: NCT04606836
Title: Analyzing the Efficacy of Peri-operative Intercostal Nerve Blocks ICNB for Acute Postoperative Pain Control in Reconstructive Breast Surgery and Mammoplasty
Brief Title: ICNBs for Post-op Pain in Breast Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Christine M. Kleinert Institute for Hand and Microsurgery (Other)
Collaborators: Jewish Hospital and St. Mary's Healthcare (Other); Baptist Health (Unknown); Kleinert, Kutz and Associates (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20.0781
Record Dates: First submitted 2020-10-12; First posted 2020-10-28 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Pain, Postoperative; Length of Stay
Keywords: ICNB; pain
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Cases will be recruited prospectively and controls will be taken retrospectively
Who Masked: Participant, Outcomes Assessor
Masking Description: The statistician will be masked to the groups the participants fall in (case vs control).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Prospective Cases (Experimental): These cases will be recruited prospectively, and receive the intercostal nerve block(s) on operated site(s). Peri-operative injections of 30 ml of 0.25% Bupivacaine each, injected over the 4th, 5th, and 6th ribs on the operated site(s).
  Interventions: Drug: Bupivacaine Hydrochloride
- Retrospective Controls (No Intervention): Controls will be gathered retrospectively from chart reviews where patient did not receive a intercostal nerve blocker bilaterally.

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — See group descriptions
  Other Names: Marcaine
  Arms: Prospective Cases

SUMMARY:
The authors will conduct this study to analyze the effectiveness of peri-operative intercostal nerve blocks (ICNBs) in reducing acute postoperative pain after reconstructive breast surgery and mammoplasty and how it affects the length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Classification (ASA Class) 3 and below.
* Bilateral or unilateral breast surgery including cancer extirpation, reconstruction (implant and expander), oncoplastic surgery (<200 gm), breast augmentation and breast reduction, etc.

Exclusion Criteria:

* Patients who refuse local anesthesia.
* Patients who cannot receive local anesthesia.
* Below the age of 20 and above the age of 70.
* Patients requiring reoperation due to complications of mammoplasty or another breast surgery.
* Poorly controlled diabetics, uncontrolled hypertension, heart disease, arrhythmias, diagnosed with bipolar and generalized anxiety disorders.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | Immediately post-operation
  Visual Analog Score (VAS) for pain compared between cases and controls, pain score on scale from 0 (no pain) to 10 (worst pain)
Post-operative pain | 30 minutes post-operation
  Visual Analog Score (VAS) for pain compared between cases and controls, pain score on scale from 0 (no pain) to 10 (worst pain)
Post-operative pain | 60 minutes post-operation
  Visual Analog Score (VAS) for pain compared between cases and controls, pain score on scale from 0 (no pain) to 10 (worst pain)
Post-operative pain | 120 minutes post-operation
  Visual Analog Score (VAS) for pain compared between cases and controls, pain score on scale from 0 (no pain) to 10 (worst pain)

SECONDARY OUTCOMES:
Length of Hospital Stay | Through study completion, average of 1 day
  time of discharge compared with time of surgery completion; Measured in number of days spent in hospital, i.e., 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Palazzo, MD, Principal Investigator — Christine M. Kleinert Institute for Hand and Microsurgery
Locations (5):
- United States (5):
  - Ambulatory Surgery Center, Kleinert Kutz Hand Care Center, New Albany, Indiana
  - Baptist Health Floyd, New Albany, Indiana
  - Christine M Kleinert Institute for Hand and Microsurgery, Louisville, Kentucky
  - HCCOC, Jewish Hospital, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky

IPD SHARING:
Plan to Share IPD: No
Only those researchers involved with the trial will have access to the individual participant data

REFERENCES:
- [Result] Park JW, Kim JH, Woo KJ. Intraoperative Intercostal Nerve Block for Postoperative Pain Control in Pre-Pectoral versus Subpectoral Direct-to-Implant Breast Reconstruction: A Retrospective Study. Medicina (Kaunas). 2020 Jun 30;56(7):325. doi: 10.3390/medicina56070325. PMID 32629834